## Prospective Randomized Evaluation of the Denali and Option Inferior Vena Cava Filters ODEN Trial: Option vs. Denali IVC Filters

## NCT02201277

Principal Investigator

Maureen P. Kohi, MD

Associate Professor of Clinical Radiology

Department of Radiology and Biomedical Imaging

Division of Vascular and Interventional Radiology

University of California, San Francisco

505 Parnassus Avenue, M-361

San Francisco, CA 94143

References from Protocol Version 1.4: March 23, 2015

## ODEN Trial References NCT02201277 – M. Kohi

- 1. Hyers TM, Agnelli G, Hull RD, et al. Antithrombotic therapy for venous thromboembolic disease. Chest 2001; 119(suppl):176S–193S.
- 2. Kinney TB. Update on inferior vena cava filters. J Vasc Interv Radiol 2003; 14:425–440.
- 3. Joels CS, Sing RF, Heniford BT. Complications of inferior vena cava filters. Am Surg 2003; 69:654–659.
- 4. Angel LF, Tapson V, Galgon RE, Restrepo MI, Kaufman J. Systematic review of the use of retrievable inferior vena cava filters. J Vasc Interv Radiol 2011; 22:1522–1530.
- 5. Decousus H, Leizorovicz A, Parent F, et al. A clinical trial of vena caval filters in the prevention of pulmonary embolism in patients with proximal deep-vein thrombosis. Prevention du Risque d'Embolie Pulmonaire par Interruption Cave Study Group. N Engl J Med 1998; 338:409–415.
- 6. Eight-year follow-up of patients with permanent vena cava filters in the prevention of pulmonary embolism: the PREPIC (Prevention du Risque d'Embolie Pulmonaire par Interruption Cave) randomized study. Circulation 2005; 112:416–422.
- 7. Ota S, Yamada N, Tsuji A, et al. The Gunther-Tulip retrievable IVC filter: clinical experience in 118 consecutive patients. Circ J 2008; 72:287–292.
- 8. Sangwaiya MJ, Marentis TC, Walker TG, Stecker M, Wicky ST, Kalva SP. Safety and effectiveness of the Celect inferior vena cava filter: preliminary results. J Vasc Interv Radiol 2009; 20:1188–1192.
- 9. Durack JC, Westphalen AC, Kekulawela S, et al. Perforation of the IVC: rule rather than exception after longer indwelling times for the Gunther Tulip and Celect retrievable filters. Cardiovasc Intervent Radiol 2012; 35: 299–308.
- 10. Kalva SP, Athanasoulis CA, Fan CM, et al. "Recovery" vena cava filter: experience in 96 patients. Cardiovasc Intervent Radiol 2006; 29:559–564.
- 11. Oliva VL, Perreault P, Giroux MF, Bouchard L, Therasse E, Soulez G. Recovery G2 inferior vena cava filter: technical success and safety of retrieval. J Vasc Interv Radiol 2008; 19:884–889.
- 12. Johnson MS, Nemcek AA Jr, Benenati JF, et al. The safety and effectiveness of the retrievable option inferior vena cava filter: a United States prospective multicenter clinical study. J Vasc Interv Radiol 2010; 21:1173–1184.

- 13. Grassi CJ, Swan TL, Cardella JF, et al. Quality improvement guidelines for percutaneous permanent inferior vena cava filter placement for the prevention of pulmonary embolism. J Vasc Interv Radiol 2003; 14(suppl): S271–S275.
- 14. Mission JF, Kerlan RK, Tan JH, Fang MC. Rates and predictors of plans for inferior vena cava filter retrieval in hospitalized patients. J Gen Intern Med 2010; 25:321–325.
- 15. Dabbagh O, Nagam N, Chitima-Matsiga R, Bearelly S, Bearelly D. Retrievable inferior vena cava filters are not getting retrieved. Where is the gap? Thromb Res 2010; 126:493–497.
- 16. Vena Caval Filter Consensus Conference. Recommended reporting standards for vena caval filter placement and patient follow-up. J Vasc Interv Radiol 2003; 14(suppl):S427–S432.
- 17. Malgor RD, Labropoulos N. A systematic review of symptomatic duode- nal perforation by inferior vena cava filters. J Vasc Surg 2012; 55:856–861.
- 18. Bogue CO, John PR, Connolly BL, Rea DJ, Amaral JG. Symptomatic caval penetration by a Celect inferior vena cava filter. Pediatr Radiol 2009; 39:1110–1113.
- 19. Wang W, Spain J, Tam MD. Acute abdominal pain after retrievable inferior vena cava filter insertion: case report of caval perforation by an Option filter. Cardiovasc Intervent Radiol 2011; 34:883–885.
- 20. Woodward EB, Farber A, Wagner WH, et al. Delayed retroperitoneal arterial hemorrhage after inferior vena cava (IVC) filter insertion: case report and literature review of caval perforations by IVC filters. Ann Vasc Surg 2002; 16:193–196.
- 21. Chintalapudi UB, Gutierrez OH, Azodo MV. Greenfield filter caval perforation causing an aortic mural thrombus and femoral artery occlusion. Cathet Cardiovasc Diagn 1997; 41:53–55.
- 22. Morishita H, Yamagami T, Matsumoto T, Takeuchi Y, Sato O, Nishimura T. Endovascular repair of a perforation of the vena caval wall caused by the retrieval of a Gunther Tulip filter after long-term implantation. Cardiovasc Intervent Radiol 2011; 34(suppl):S321–S323.
- 23. Ford ME, Lippert JA, McGraw K. Symptomatic Filter Penetration Presenting as Pancreatitis. J Vasc Interv Radiol 2010; 21:574–576.
- 24. Caplin DM, Nikolic B, Kalva SP, Ganguli S, Saad WE, Zuckerman DA. Quality Improvement Guidelines for the Performance of Inferior Vena Cava Filter Placement for the Prevention of Pulmonary Embolism. J Vasc Interv Radiol 2011; 22:1499–1506
- 25. Olorunsola OG, Kohi MP, Fidelman N, Westphalen AC, Kolli KP, Taylor AG, Gordon RL, LaBerge JM, Kerlan RK. Caval Penetration by Retrievable Inferior Vena Cava Filters: A Retrospective Comparison of Option and Gunther-Tulip Filters. J Vasc Interv Radiol 2013; 24:566–571.
- 26. Durack JC, Westphalen AC, Kekulawela S, Bhanu SB, Avrin DE, Gordon RL, Kerlan RK.

- Perforation of the IVC: Rule Rather Than Exception After Longer Indwelling Times for the Gunther Tulip and Celect Retrievable Filters. Cardiovasc Intervent Radiol (2012) 35:299–308.
- 27. Zhou D, Spain J,Moon E, Mclennan G, Sands MJ, Wang W. Retrospective Review of 120 Celect Inferior Vena Cava Filter Retrievals: Experience at a Single Institution. J Vasc Interv Radiol 2012; 23:1557–1563
- 28. Stein PD, Kayali F, Olson RE. Twenty-one-year trends in the use of inferior vena cava filters. Arch Intern Med 2004164(14):1541–1545.
- 29. Jaff MR, Goldhaber SZ, Tapson VF. High utilization rate of vena cava filters in deep vein thrombosis. Thromb Haemost 2005 93:1117–1119.
- 30. Athanasoulis CA, Kaufman JA, Halpern EF et al. Inferior vena cava filters: review of a 26-year single-center clinical experience. Radiology 2000 216:54–66.
- 31. Ray CE, Mitchell E, Zipser S et al.Outcomes with retrievable inferior vena cava filters: a multicenter study. J Vasc Interv Radiol 200617:1595–1604.
- 32. Karmy-Jones R, Jurkovich GJ, Velmahos GC et al. Practice patterns and outcomes of retrievable vena cava filters in trauma patients: an AAST multicenter study. J Trauma 2007 62:17–24
- 33. White RH, Zhou H, Kim J et al. A population-based study of the effectiveness of inferior vena cava filter use among patients with venous thromboembolism. Arch Intern Med 2000 160:2033–2041.
- 34. Girard P, Stern J, Parent F. Medical literature and vena cava filters: so far so weak. Chest 2002 122(3):963–967.
- 35. Ray CE, Kaufman JA. Complications of inferior vena cava filters. Abdom Imaging 1996 21(4):368–374.
- 36. Greenfield L, Proctor M. Filter complications and their management. Semin Vasc Surg 2000 13:213–216.
- 37. Sadaf A, Rasuli P, Olivier A et al. Significant caval penetration by the Celect inferior vena cava filter: attributable to filter design? J Vasc Interv Radiol 200718(11):1447–1450.
- 38. Dardik A, Campbell KA, Yeo CJ et al. Vena cava filter ensnarement and delayed migration: an unusual series of cases. J Vasc Surg 1997 26:869–874.
- 39. Smouse HB, Van Alstine WG, Mack S et al. Deployment performance and retrievability of the Cook Celect vena cava filter. J Vasc Interv Radiol 2009 20:375–383.

- 40. Goldman HB, Hanna K, Dmochowski RR. Ureteral injury secondary to an inferior vena caval filter. J Urol 1996 156:1763.
- 41. Sarkar MR, Lemminger FM. An unusual case of upper gastrointestinal hemorrhage—perforation of a vena cava filter into the duodenum. Vasa 1997 26:305–307.

## Retrieval:

- 42. Turba UC, Arslan B, Meuse M et al (2010) Gunter tulip filter retrieval experience: predictors of successful retrieval. Cardiovasc Intervent Radiol 2010 33:732–738.
- 43. Mission JF, Kerlan RK Jr, Tan JH et al. Rates and predictors of plans for inferior vena cava filter retrieval in hospitalized patients. J Gen Intern Med 2010 25(4):321–325.
- 44. Kuo WT, Cupp JS, Louie JD et al. Retrieval of permanently-embedded IVC filters and description of the laser-assisted sheath technique: radiographic-histopathologic correlation. J Vasc Interv Radiol Suppl 2010 21(2):4.
- 45. Stavropoulos SW, Dixon RG, Burke CT et al. Embedded inferior vena cava filter removal: use of endobronchial forceps. J Vasc Interv Radiol 2008 19:1297–1301.
- 46. Rubenstein L, Chun AK, Chew M et al. Loop-snare technique for difficult inferior vena cava filter retrievals. J Vasc Interv Radiol 2007 18:1315–1318.
- 47. Kuo WT, Bostaph AS, Loh CT et al. Retrieval of trapped Gunther Tulip inferior vena cava filters: snare-over-guide wire loop technique. J Vasc Interv Radiol 2006 17:1845–1849.
- 48. Food and Drug Administration. <u>"Inferior Vena Cava (IVC) Filters: initial Communication: Risk of Adverse Events with Long Term Usage"</u>. United States Food and Drug Administration. Retrieved 2010-09-09.